CLINICAL TRIAL: NCT00324623
Title: Phase I Study of In Vivo Expansion of Melan-A/MART-1 Antigen-Specific CD8 T Lymphocytes Following Transient Immunosuppression in Patients With Advanced Melanoma
Brief Title: Cyclophosphamide and Fludarabine Followed by Cellular Adoptive Immunotherapy and Vaccine Therapy in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Serge Leyvraz (Other)
Responsible Party: Sponsor-Investigator, Prof. Serge Leyvraz, Chef de Service, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000468827; CHUV-CEPO-ITA-02; EU-20607
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Immunotherapy, Adoptive; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphodepletion, vaccine, IMP321 adjuvant (Experimental)
  Interventions: Biological: Melan-A VLP vaccine, IMP321 adjuvant; Biological: adoptive immunotherapy; Biological: therapeutic autologous lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: Melan-A VLP vaccine, IMP321 adjuvant
Biological: adoptive immunotherapy
Biological: therapeutic autologous lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide and fludarabine, may be used to prepare the body for other treatments, such as cellular adoptive immunotherapy. Biological therapies, such as cellular adoptive immunotherapy, may stimulate the immune system in different ways and stop tumor cells from growing. Vaccines may help the body build an effective immune response to kill tumor cells. Giving cyclophosphamide together with fludarabine followed by biological therapy may be an effective treatment for metastatic melanoma.

PURPOSE: This phase I trial is studying the side effects of giving cyclophosphamide together with fludarabine followed by cellular adoptive immunotherapy, and vaccine therapy in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the magnitude and duration of the expansion of antigen-specific T-cells present in post-vaccination peripheral blood mononuclear cells and reinfused after immunosuppression in patients with metastatic melanoma.
* Characterize the T-cell subsets (phenotype, function, T-cell receptor repertoire) in these patients.
* Determine the tumor response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label dose-finding study. Patients undergo leukapheresis to collect whole peripheral blood mononuclear cells (PBMC). Patients are then assigned to 1 of 3 treatment groups.

* Group 1 (closed to accrual as of 5/8/2007): Patients receive cyclophosphamide IV on days -7 and -6 and fludarabine IV on days -5 to -3. Patients undergo autologous PBMC infusion on day 0. Patients also receive vaccination comprising Melan-A vaccine emulsified in incomplete Freund's adjuvant (IFA) subcutaneously (SC) once every 3 weeks beginning on day 0.
* Group 2 (closed to accrual as of 8/15/2007): Patients receive cyclophosphamide IV at a higher dose than in group 1 on days -7 and -6 and fludarabine IV on days -5 to -3. Patients also receive an autologous PBMC infusion and Melan-A vaccine emulsified in IFA as in group 1.
* Group 3: Patients receive cyclophosphamide IV at 30 mg/kg on days -7 and -6. Patients also receive fludarabine 30 mg/m2 IV on days -5 to -3, autologous PBMC infusion on day 0,and Melan-A vaccine emulsified in IFA and IMP321. The first 3 patients receive 25 micrograms of IMP321, in the absence of severe 3 or 4 toxicity, the dose will be escalated to IMP321 250 micrograms.

PROJECTED ACCRUAL: A total of 9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma
* Progressive disease after receiving prior Melan-A peptide vaccine on an immunotherapy protocol of the Ludwig Institute AND achieved a detectable immune response (increase of specific CD8^+ TET^+ Melan-A)
* Tumor must express MART-1/Melan-A antigen
* HLA-A2 positive
* Not eligible for other protocols due to progressive disease OR maximum number of vaccine injections with stable disease has been attained

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Whole blood counts normal
* Pulmonary status normal
* Transaminases < 1.5 times upper limit of normal (ULN)
* Gamma-glutamyl-transferase < 1.5 times ULN
* Bilirubin normal
* Creatinine clearance > 70 mL/min
* No major uncontrolled heart disease
* No arterial hypertension

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior chemotherapy, biologic therapy, radiotherapy, and/or surgery allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-09; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Phenotype, function, and T-cell receptor repertoire | Anti-tumor immune response evaluated at each vaccine and until the last administered vaccine
Tumor response | Tumor response evaluated 4 weeks after last vaccine
Toxicity | Within 30 days after completion of the last vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Serge Leyvraz, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Romano E, Michielin O, Voelter V, Laurent J, Bichat H, Stravodimou A, Romero P, Speiser DE, Triebel F, Leyvraz S, Harari A. MART-1 peptide vaccination plus IMP321 (LAG-3Ig fusion protein) in patients receiving autologous PBMCs after lymphodepletion: results of a Phase I trial. J Transl Med. 2014 Apr 12;12:97. doi: 10.1186/1479-5876-12-97. PMID 24726012